CLINICAL TRIAL: NCT01255085
Title: The Effect of Yellow Pea Protein and Fiber on Short Term Food Intake, Subjective Appetite and Glycemic Response in Healthy Young Males
Brief Title: Yellow Pea Protein and Fibre and Short Term Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PureNet_22627
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Type II Diabetes Mellitus; Metabolic Syndrome
Keywords: Obesity; Food intake regulation; blood glucose regulation; protein; fiber; pulses; yellow peas
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- 10 g of yellow pea fiber (Experimental)
  Interventions: Dietary Supplement: yellow pea fiber
- 20 g of yellow pea fiber (Experimental)
  Interventions: Dietary Supplement: yellow pea fiber
- 10 g of yellow pea protein (Experimental)
  Interventions: Dietary Supplement: yellow pea protein
- 20 g of yellow pea protein (Experimental)
  Interventions: Dietary Supplement: yellow pea protein
- Control Tomato Soup (Experimental)
  Interventions: Dietary Supplement: Control Tomato Soup

INTERVENTIONS:
Dietary Supplement: yellow pea protein — Served in a tomato soup
  Arms: 10 g of yellow pea protein; 20 g of yellow pea protein
Dietary Supplement: yellow pea fiber — Served in a tomato soup
  Arms: 10 g of yellow pea fiber; 20 g of yellow pea fiber
Dietary Supplement: Control Tomato Soup — Served in a tomato soup
  Arms: Control Tomato Soup

SUMMARY:
It is hypothesized that yellow pea protein and fiber will reduce short-term food intake, subjective appetite and glycemic response.

DETAILED DESCRIPTION:
A within-subject, randomized study was conducted. Each subject returned 5 times, 1 week apart, and received 1 of the 5 treatments per week. The 5 treatments were tomato soup with 10 or 20 g of isolated yellow pea fibre or protein, or a control soup with no added pea fractions. Food intake was measured at an ad libitum pizza meal served 30 minutes after treatment. Satiety and blood glucose (via finger prick) were measured throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* male 20-30 years old healthy weight

Exclusion Criteria:

* smoking restrictive eating metabolic diseases breakfast skippers dieters

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Energy Intake | at 30 minutes after treatment
  Energy intake at an ad libitum pizza meal

SECONDARY OUTCOMES:
Glycemic Response | 0-170 minutes post treatment
  Blood Glucose every 15-30 minutes via finger prick
Subjective Appetite | 0-170 minutes post treatment
  Subjective Appetite measured every 15-30 minutes via Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto - Department of Nutritional Sciences, Toronto, Ontario, Canada